CLINICAL TRIAL: NCT02285933
Title: Does the Addition of Virtual Reality Training to a Standard Program of Inpatient Rehabilitation Improve Sitting Balance Ability and Function After Stroke? A Blinded Randomized Controlled Trial.
Brief Title: Virtual Reality Exercise for Stroke Rehabilitation in Inpatients Who Are Unable to Stand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Ottawa Hospital Research Institute (Other); University of Ottawa (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Hillel Finestone, Director of Stroke Rehabilitation Research, Bruyère Health Research Institute.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-14-0005830
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: stroke; physical therapy specialty; exercise therapy; virtual reality; man-machine systems; randomized control trial; inpatients; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRT (Experimental): sitting balance exercises delivered via virtual reality training
  Interventions: Other: virtual reality training
- control (Active Comparator): virtual reality training requiring limited arm movements and no challenge to sitting balance
  Interventions: Other: control

INTERVENTIONS:
Other: virtual reality training — Each participant will engage in 10-12 sessions of 30-50 minutes each of virtual reality training (VRT) using Jintronix Rehabilitation Software and three-dimensional motion capture technology. A camera captures the movements of the participant and allows him or her to control an avatar, which interacts with the game. Exercises challenge sitting balance control, reaching and shifting the base of support; for example, controlling a ball as it rolls down a maze or reaching to put dishes away in a virtual kitchen. The difficulty of the games is monitored to maintain a challenge to sitting balance. The participant sits on a CONFORMat pressure mat which continuously monitors his or her centre of pressure to ensure that the participant is adequately challenged during the VRT.
  Arms: VRT
Other: control — Each participant will engage in 10-12 sessions of 30-50 minutes each of virtual reality training (VRT) using Jintronix Rehabilitation Software and three-dimensional motion capture technology. A camera captures the movements of the participant and allows him or her to control an avatar, which interacts with the game. Control group exercises require limited hand and arm movements; for example, using an arm to move a fish along a simple pathway or using the arms to pop balloons without reaching. Control group participants are strapped into their chair to minimize trunk movement. The participant sits on a CONFORMat pressure mat which continuously monitors his or her centre during the VRT.
  Arms: control

SUMMARY:
The purpose of this study is to determine if the addition of 10 to 12 sessions of sitting balance exercises using virtual reality training will provide additional gains in balance ability and function over standard inpatient rehabilitation in stroke patients.

DETAILED DESCRIPTION:
Introduction Sitting balance may be affected by stroke, resulting in functional impairment and reduced mobility. Early return of sitting balance predicts greater return of motor function and mobility after stroke. Task-specific therapy is effective but patients must be motivated to perform the exercises repeatedly for the greatest benefit.

Virtual reality training (VRT) allows patients to do exercises while interacting with a video game interface. It is enjoyable and may encourage repetition of therapeutic exercises. Past work in our laboratory showed that standing balance exercises performed with VRT produced additional improvements in gait speed and leg function over traditional inpatient rehabilitation (1). Because of legislative change in Ontario most stroke rehabilitation inpatients today cannot stand independently. There have been no studies on the effect of VRT on sitting balance.

Purpose To assess whether additional sitting balance exercises performed via VRT can improve sitting balance and sitting function (ex. reaching) in stroke rehabilitation inpatients.

Hypothesis The addition of VRT for sitting balance will significantly improve sitting balance and function, beyond the gains realized from traditional inpatient rehabilitation.

Experimental Approach In this blinded randomized control trial funded by the Heart & Stroke Foundation, 76 participants with stroke will be recruited from an inpatient rehabilitation unit. This number will provide enough power to detect a large effect size (0.83) with the primary outcome measure and accounting for a 20% drop-out rate. Individuals who are medically stable and who can sit for at least 20 minutes with or without trunk support but cannot stand independently for more than one minute will be eligible. These criteria will target our selection to those who need to work most on sitting balance. Participants will be randomized into experimental and control groups.

Participants in both groups will perform VRT for 30-50 minutes daily for 10-12 sessions, in addition to their rehabilitation program. VRT will be delivered with Jintronix software and motion capture technology. Exercises for the experimental group will challenge sitting balance control, reaching and shifting the base of support. Control group exercises will require limited hand and arm movements, to equalize the additional time spent in an engaging activity without working on trunk balance. Control group participants will be strapped into their chair to minimize trunk movement. A CONFORMat pressure mat will be used to monitor centre of pressure changes during the intervention.

Outcome measures will be performed pre-, post- and 1 month post-intervention, by an assessor blinded to group allocation. The primary outcome measure will be the Function in Sitting Test. Secondary outcome measures will be: Ottawa Sitting Scale, Reaching Performance Scale, Wolf Motor Function Test and quantitative measures of postural control performed in sitting. Two-way analyses of variance [factors: time (pre-, post-, 1 month post-)and group(experimental, control)] and Tukey's post-hoc analyses will be used to test the effect of VRT on the outcome measures.

Significance and Knowledge Translation If we show that the addition of sitting balance exercises via VRT to traditional rehabilitation improves sitting balance and function, VRT may be added to inpatients' rehabilitation therapy. The ultimate goal is to improve the quality of patients' lives and decrease the burden on their caregivers. Since the Jintronix system is portable, we hope to acquire funding for several units. We would then be able to assess the use of VRT by therapists for inpatients and outpatients with stroke.

(1) McEwen D et al. Stroke 2014;45:1853-1855

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke in the left or right cortical or subcortical regions
* medically stable
* cannot stand independently for >1 minute or cannot stand at all
* can sit for at least 20 minutes with or without trunk support and can sit for at least 1 minute without trunk support
* able to provide informed consent

Exclusion Criteria:

* unstable cardiovascular, respiratory, endocrine, orthopedic or neurological condition that precludes exercise of low to moderate intensity
* vestibular deficits or vertigo
* seizure activity in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the Function In Sitting Test (FIST) from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses static, dynamic and reactional sitting balance
Change in the Function In Sitting Test (FIST) from baseline to 1 month after second assessment | baseline,1 month after second assessment
  assesses static, dynamic and reactional sitting balance

SECONDARY OUTCOMES:
Change in the Ottawa Sitting Scale (OSS) from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses static and dynamic sitting balance
Change in the Ottawa Sitting Scale (OSS) from baseline to 1 month after second assessment | baseline, 1 month after second assement
  assesses static and dynamic sitting balance
Change in Limits of stability in sitting (LoS) from baseline to after 10-12 treatment sessions | before treatment, immediately after 10-12 treatments
  assesses dynamic sitting balance using a force plate or pressure mat
Change in Limits of stability in sitting (LoS) from baseline to 1 month after second assessment | baseline, 1 month after second assement
  assesses dynamic sitting balance using a force plate or pressure mat
Change in Postural sway in sitting from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses static sitting balance using a force plate or pressure mat
Change in Postural sway in sitting from baseline to 1 month after second assessment | baseline, 1 month after second assement
  assesses static sitting balance using a force plate or pressure mat
Change in the Reaching Performance Scale (RPS) from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses sitting balance function during reaching
Change in the Reaching Performance Scale (RPS) from baseline to 1 month after second assessment | baseline, 1 month after second assement
  assesses sitting balance function during reaching
Change in the Wolf Motor Function Test (WMFT) from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses sitting balance function using global arm function
Change in the Wolf Motor Function Test (WMFT) from baseline to 1 month after second assessment | baseline, 1 month after second assement
  assesses sitting balance function using global arm function
Change in The Motivation for Physical Activity Questionnaire from baseline to after 10-12 treatment sessions | before treatment, immediately after 10-12 treatments
  Likert scale from 0-6 to assess motivation to engage in exercise
Change in The Motivation for Physical Activity Questionnaire from baseline to 1 month after second assessment | baseline, 1 month after second assement
  Likert scale from 0-6 to assess motivation to engage in exercise
Change in the Behavioral Regulation in Exercise Questionnaire (BREQ-2) from baseline to after 10-12 treatment sessions | baseline, immediately after 10-12 treatments
  assesses quality of motivation to engage in exercise
Change in the Behavioral Regulation in Exercise Questionnaire (BREQ-2) from baseline to 1 month after second assessment | baseline, 1 month after second assessment
  assesses quality of motivation to engage in exercise
Psychosocial Impact of Assistive Devices Scale (PIADS) | immediately after 10-12 treatments
  assesses the psychosocial impact of assistive devices or technology on "functional independence, well-being and quality of life"
Psychosocial Impact of Assistive Devices Scale (PIADS) | 1 month after first assement
  assesses the psychosocial impact of assistive devices or technology on "functional independence, well-being and quality of life"
The ability to enroll an average of five new participants a month, to obtain a consent rate of 60% of eligible patients and a rate of protocol violations resulting in noncompliance with VRT of less than 10%. | immediately after 76 participants have finished the protocol and assessments
  assesses the feasibility of performing a larger multicentre trial of VRT with rehabilitation inpatients

CONTACTS AND LOCATIONS:
Overall Officials: Hillel M Finestone, MD, Principal Investigator — Bruyère Health Research Institute.; Heidi Sveistrup, PhD, Study Director — University of Ottawa; Martin Bilodeau, PhD, Study Director — University of Ottawa
Locations (1):
- Elisabeth Bruyere Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
As this is not part of a larger, multi-centre trial, we do not plan to share our data.

REFERENCES:
- [Background] McEwen D, Taillon-Hobson A, Bilodeau M, Sveistrup H, Finestone H. Virtual reality exercise improves mobility after stroke: an inpatient randomized controlled trial. Stroke. 2014 Jun;45(6):1853-5. doi: 10.1161/STROKEAHA.114.005362. Epub 2014 Apr 24. PMID 24763929
- [Background] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Fergusson D, Levac D, Finestone H. Does the addition of virtual reality training to a standard program of inpatient rehabilitation improve sitting balance ability and function after stroke? Protocol for a single-blind randomized controlled trial. BMC Neurol. 2016 Mar 31;16:42. doi: 10.1186/s12883-016-0563-x. PMID 27036515
- [Derived] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Finestone H. Implementation of a randomized controlled trial on an inpatient stroke rehabilitation unit: Lessons learned. Contemp Clin Trials Commun. 2020 Apr 6;18:100563. doi: 10.1016/j.conctc.2020.100563. eCollection 2020 Jun. PMID 32617429
- [Derived] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Yang C, Finestone H. Sitting Balance Exercise Performed Using Virtual Reality Training on a Stroke Rehabilitation Inpatient Service: A Randomized Controlled Study. PM R. 2020 Aug;12(8):754-765. doi: 10.1002/pmrj.12331. Epub 2020 Feb 21. PMID 31970898